CLINICAL TRIAL: NCT05747131
Title: Unified Protocol for Transdiagnostic Treatment of Emotional Disorders in Children: A Multicenter Study to Assess the Acceptability, Feasibility and Efficacy of a Blended Format of the Program in Portugal
Brief Title: Emotion Detectives In-Out: Feasibility and Efficacy of a Blended Version of the Unified Protocol for Children
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Coimbra (Other)
Collaborators: Fundação para a Ciência e a Tecnologia (Other); University of Lisbon (Other)
Responsible Party: Principal Investigator, Helena Moreira, Prof., University of Coimbra
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PTDC/PSI-GER/0689/2020
Record Dates: First submitted 2023-02-07; First posted 2023-02-28 (Actual); Last update posted 2023-05-12 (Actual); Status verified 2023-05

CONDITIONS: Anxiety Disorders
Keywords: Unified Protocol; Children; Blended therapy; Parents
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Emotion Detectives In-Out (Experimental): Emotion Detectives In-Out consists of 15 weekly sessions with the children (9 face-to-face group sessions, 4 online sessions and 2 videoconference sessions).
  Interventions: Behavioral: Emotion Detectives In-Out
- Coping Cat (Active Comparator): Coping Cat consists of 16 weekly group sessions with the children (5 to 7 children per group) and 2 sessions with the parents.
  Interventions: Behavioral: Coping Cat

INTERVENTIONS:
Behavioral: Emotion Detectives In-Out — Emotion Detectives In-Out is a blended cognitive-behavioral intervention for children with emotional disorders aged between 7 to 12 years and their parents. It contains group sessions, online self-guided sessions and videoconference sessions. The groups will consist of about 5 to 7 children. Face-to-face sessions have an expected duration of 90 minutes and will be implemented by clinical psychologists with specific training in the program. The online sessions were developed by the research team and are completely self-guided. These sessions last approximately 45 minutes. Parents will be asked to participate in 2 face-to-face sessions, 4 videoconference sessions and 10 self-guided online sessions. It is a transdiagnostic and emotion-focused manualized cognitive-behavioral therapy designed to help children reduce the intensity and frequency of strong and aversive emotional experiences and to help parents reduce parental emotional behaviors.
  Arms: Emotion Detectives In-Out
Behavioral: Coping Cat — Coping Cat is a cognitive behavioral therapy for children with anxiety aged between 7 to 13 years. Coping Cat consists of 16 weekly group sessions with the children (5 to 7 children per group) and 2 sessions with the parents. Face-to-face sessions have an expected duration of 90 minutes and will be implemented by clinical psychologists.
  Arms: Coping Cat

SUMMARY:
The goal of this clinical trial is to test the efficacy of a blended format (i.e., a combination of face-to-face and online sessions into one integrated treatment protocol) of the Unified Protocol for Transdiagnostic Treatment of Emotional Disorders in Children (UP-C) in a sample of children aged between 7 and 12 years with a primary diagnosis of an anxiety disorder or with clinically significant levels of anxiety.

The main questions it aims to answer are:

* Is the proposed intervention (named Emotion Detectives In-Out) feasible and acceptable among Portuguese children with anxiety disorders and their parents?
* Is the Emotion Detectives In-Out intervention as effective as an evidence-based intervention for children's anxiety disorders in reducing anxiety symptomatology and changing secondary outcomes?
* What are the key predictors of adherence to the Emotion Detectives In-Out intervention?
* What are the key predictors of treatment outcomes?

Participants (children and one parent/legal representative) will:

* Participate in an initial interview with a clinical psychologist, who will assess if children and parents meet eligibility criteria.
* Complete an assessment protocol before, during, and after the intervention, as well as three months later.
* Be randomly assigned to one of the two conditions: experimental (Emotion Detectives In-Out) or active control (Coping Cat).
* Participate in one of the two psychological interventions. Researchers will compare the experimental and control groups to see if the Emotion Detectives In-Out intervention is equally efficacious as the Coping Cat intervention.

DETAILED DESCRIPTION:
Childhood emotional disorders, particularly anxiety disorders, are an important public health concern due to their high and increasing prevalence, impact on children's functioning in multiple domains (e.g., family, academic, social), and long-term consequences. However, there is a significant gap between their needs and access to mental healthcare, with most children lacking access to evidence-based treatments (EBT). Several factors can contribute to a lack of adequate mental health care for children, including an insufficient number of trained clinicians, the difficulty of effectively disseminating the multitude of disorder-specific EBTs for emotional disorders to clinicians, and other barriers to face-to-face treatment. An Internet-based intervention can be an effective solution to overcome these difficulties. This project aims to develop and test the efficacy of a blended intervention of the Unified Protocol for Transdiagnostic Treatment of Emotional Disorders in Children (UP-C).

The UP-C is a cognitive-behavioral therapy (CBT) that takes a transdiagnostic approach to treating multiple emotional disorders simultaneously by addressing shared mechanisms underlying these disorders and employing a common set of EBT strategies (e.g., exposure, mindfulness). It is a child-friendly extension of the adult UP that delivers the UP core components in an interactive and child-friendly group format with extensive parent involvement. It has 15 weekly sessions for children and 15 weekly sessions for parents with an approximate duration of 90 minutes each. With a blended approach the researchers aim to improve the delivery of UP-C, by retaining the benefits of face-to-face and online therapy, while mitigating their limitations. This new version is expected to reduce costs of the therapy for families and institutions while also increasing compliance, motivation, uptake of treatment principles, and facilitating generalization of the application of core treatment components.

The blended version of the UP-C, named "Emotion Detectives In-Out" consists of 15 weekly sessions with the children (9 face-to-face group sessions, 4 online self-guided sessions and 2 videoconference sessions). The groups will consist of about 5 to 7 children. Face-to-face sessions have an expected duration of 90 minutes and will be implemented by clinical psychologists with specific training in the program. The online sessions were developed by the research team and are completely self-guided. These sessions last approximately 45 minutes. Parents will be asked to participate in 2 face-to-face sessions, 4 videoconference sessions and 10 self-guided online sessions.

ELIGIBILITY:
Inclusion Criteria:

1. The child is aged between 7 and 12 years;
2. The child has a primary diagnosis of an anxiety disorder or clinically significant anxiety symptoms;
3. Both the child and the parent are able to speak, read and understand Portuguese;
4. Both the child and the parent have Internet access.

Exclusion Criteria:

1. Diagnosis of a psychotic disorder, bipolar disorder, intellectual disability or autism spectrum disorder;
2. Severe current suicidal ideation;
3. The child is not on a stable dose of a psychotropic or other type of medication for at least 1 month prior to T0 assessment;
4. The child has previously received CBT with exposure techniques.

Ages: 7 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 180 (Estimated)
Dates: Start 2023-09 (Estimated); Primary Completion 2024-07 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Change in anxiety symptoms as measured by the Revised Children's Anxiety and Depression Scale (RCADS). | Baseline, Mid-treatment (week 7), within 1 week post-treatment, 3 months follow-up]
  The Revised Children's Anxiety and Depression Scale is a 47 item self-report questionnaire that measures symptoms of depression and anxiety in children and adolescents aged 8 - 18. It has 6 subscales: separation anxiety disorder, social phobia, generalized anxiety disorder, panic disorder, obsessive compulsive disorder, and low mood (major depressive disorder). It yields a Total Anxiety Scale (the sum of the 5 anxiety subscales) and a Total Anxiety & Depression Scale (sum of all 6 subscales). The Total Anxiety Scale ranges from 0 to 111, and the Total Anxiety & Depression scale ranges from 0 to 141, with higher scores indicating increased symptom severity.
Change in anxiety symptoms as measured by the Revised Children's Anxiety and Depression Scale - Parent version (RCADS-P). | Baseline, Mid-treatment (week 7), within 1 week post-treatment, 3 months follow-up
  The Revised Child Anxiety and Depression Scale - Parent Version (RCADS-P) is a 47 item parent-reported questionnaire that measures symptoms of depression and anxiety in children and adolescents aged 8 - 18. It has 6 subscales: separation anxiety disorder, social phobia, generalized anxiety disorder, panic disorder, obsessive compulsive disorder, and low mood (major depressive disorder). It yields a Total Anxiety Scale (the sum of the 5 anxiety subscales) and a Total Anxiety & Depression Scale (sum of all 6 subscales). The Total Anxiety Scale ranges from 0 to 111, and the Total Anxiety & Depression scale ranges from 0 to 141, with higher scores indicating increased symptom severity.
Change in anxiety symptoms as measured by the Clinician Global Impression - Improvement scale (CGC-I). | within 1 week post-treatment
  Higher scores indicate increased symptom worsening.
Change in severity of anxiety symptoms as measured by the Clinician Global Impression - Severity scale (CGC-S). | Baseline, within 1 week post-treatment
  The Clinician Global Impression - Severity scale is a one-item measure assessing the clinician's perception of the severity of the patient's symptoms, with scores ranging from 1 (not at all ill) to 7 (extremely ill). Higher scores indicate increased symptom severity.

SECONDARY OUTCOMES:
Change in the interference of anxiety in child's life, as measured by the Child Anxiety Life Interference Scale - Self-Report (CALIS-C) | Baseline, Mid-treatment (week 7), within 1 week post-treatment, 3 months follow-up
  The Child Anxiety Life Interference Scale - Self-Report consists of a 9-item scale administered to children. Items are rated on a 5-point Likert scale (0 = not at all to 4 = a great deal). The total score ranges from 0 to 36, with higher scores indicating greater interference of anxiety symptoms in children's life.
Change in the interference of anxiety in child's life, as measured by the Child Anxiety Life Interference Scale - Parent's Report (CALIS-P) | Baseline, Mid-treatment (week 7), within 1 week post-treatment, 3 months follow-up
  The Child Anxiety Life Interference Scale - Parent's Report consists of two 9-item scales (Child Interference Subscale and Family Interference Subscale) administered to parents. Items are rated on a 5-point Likert scale (0 = not at all to 4 = a great deal). The total scores of the Child Interference Subscale and of the Family Interference Subscale range from 0 to 36, with higher scores indicating greater interference of anxiety symptoms in the lives of children and families, respectively.
Change in children's behavioral avoidance, as measured by the Child Avoidance Measure Self-Report (CAMS) | Baseline, Mid-treatment (week 7), within 1 week post-treatment, 3 months follow-up
  The Child Avoidance Measure Self-Report is an 8-item self-report measure that assesses children's behavioral avoidance when faced with stimuli that elicit anxiety, fear, or worry, from the child's perspective. Items are rated on a 4-point Likert scale (0 = Almost Never to 3 = Almost Always). The total score ranges from 0 to 24, with higher scores indicating higher behavioral avoidance.
Change in children's behavioral avoidance, as measured by the Child Avoidance Measure Parent-Report (CAMP) | Baseline, Mid-treatment (week 7), within 1 week post-treatment, 3 months follow-up
  The Child Avoidance Measure Parent-Report is an 8-item measure that assesses children's behavioral avoidance when faced with stimuli that elicit anxiety, fear, or worry, from the parents' perspective. Items are rated on a 4-point Likert scale (0 = Never, almost never, or not an issue to 3 = Almost Always). The total score ranges from 0 to 24, with higher scores indicating higher behavioral avoidance.
Change in children's positive and negative affect, as measured by the Positive and Negative Affect Schedule for Children - Short Version (PANAS-C-SF) | Baseline, Mid-treatment (week 7), within 1 week post-treatment, 3 months follow-up
  The Positive and Negative Affect Schedule for Children - Short Version has 10 items and is composed by two subscales (Positive Affect and Negative Affect). Items are answered in a 5-item Likert scale that ranges from 1 (Very slightly or not at all) to 5 (Extremely). Both subscales can range from 5 to 25, with higher scores on Positive Affect indicating greater intensity of positive emotions, and higher scores on Negative Affect indicating greater intensity of negative emotions.
Change in children's anxiety sensitivity, as measured by the Children's Anxiety Sensitivity Inventory-Revised (CASI-R). | Baseline, Mid-treatment (week 7), within 1 week post-treatment, 3 months follow-up
  The Children's Anxiety Sensitivity Inventory-Revised is a 31 item self-report scale that measures children's anxiety sensitivity across four domains: fear of cardiovascular symptoms, fear of publicly observable anxiety reactions, fear of cognitive dyscontrol and fear of respiratory symptoms. Items are answered in a 3-item Likert scale that ranges from 0 (Not true) to 3 (Very true). A total anxiety sensitivity score can be obtained by summing across all items and ranges from 0 to 93, with higher scores indicating higher anxiety sensitivity.
Change in children's difficulties in emotion expression, as measured by the Emotional Expression Scale for Children (EESC) | Baseline, Mid-treatment (week 7), within 1 week post-treatment, 3 months follow-up
  The Emotional Expression Scale for Children is a 16 item self-report questionnaire that assesses children's difficulties in emotion expression (i.e., poor emotion awareness and reluctance to express emotions). Items are answered on a 5-point Likert-type scale that ranges from 1 (Not at All True) to 5 (Extremely true). The total score ranges from 16 to 80, with higher scores indicating greater difficulty in expressing emotions.
Change in children's negative cognitive errors, as measured by the Children's Negative Cognitive Error Questionnaire (CNCEQ) | Baseline, Mid-treatment (week 7), within 1 week post-treatment, 3 months follow-up
  The Children's Negative Cognitive Error Questionnaire is a 24 item self-report questionnaire that assesses four types of cognitive errors: catastrophizing, overgeneralizing, personalizing, and selective abstraction. Items are answered on a 5-point scale that ranges from 1 (Nothing like I would think) to 5 (Exactly what I would think). A total cognitive distortion score can be obtained, ranging from 24 to 120. Higher scores indicate more distorted cognitive processes.
Change in children's quality of life, as measured by the KIDSCREEN-10 Index (Parent Report) | Baseline, Mid-treatment (week 7), within 1 week post-treatment, 3 months follow-up
  The KIDSCREEN-10 Index (parent report) assesses children's overall levels of quality of life (physical, mental and social) as reported by their parents. Items are answered on a 5-point Likert scale ranging from 1 (never/not at all) to 5 (always/extremely). The sum of all items provides a global index of quality of life. The standardized scores ranges from 0 to 100, with higher results suggesting a better quality of life.
Change in parental overprotection, as measured by the Parental Anxiety and Overprotection Scale (PAOS) | Baseline, within 1 week post-treatment, 3 months follow-up
  The Parental Anxiety and Overprotection Scale assesses parents' overprotection behaviors and other behaviors that aim to encourage children to cope with and face situations that cause them anxiety. The parental overprotection subscale has 7 items and the support of children's coping behaviors subscale has 3 items, which are both rated on a 5-point Likert scale ranging from 0 (nothing) to 4 (a lot). The total score of the overprotection subscale can range from 0 to 28 and total score of the support of children's coping behaviors subscale can range from 0 to 12, with higher scores indicating higher levels of parental overprotection and higher levels of parental supportive behaviors, respectively.
Change in parental criticism as measured by the Egna Minnen Beträffande Uppfostran Scale (EMBU-P) | Baseline, within 1 week post-treatment, 3 months follow-up
  The Rejection subscale of Egna Minnen Beträffande Uppfostran Scale assesses parents' levels of criticism towards their child. This subscale has 17 items answered on a 4-point Likert scale that ranges from 1 (No, never) to 4 (Yes, always). The total rejection score can range from 17 to 68, with higher scores suggesting higher levels of rejection and criticism.
Change in parental modeling of intense emotions, as measured by the Parent Emotion Regulation Scale (PERS) | Baseline, within 1 week post-treatment, 3 months follow-up
  The Parents' Lack of Emotional Control subscale of the Parent Emotion Regulation Scale assesses parents' lack of ability to modulate their own negative emotions in the presence of the child. This subscale has 4 items answered on a 5-point Likert scale that ranges from 0 (never or almost never) to 4 (always or almost always). The total score can range from 0 to 4, with higher scores indicating a higher level of negative emotion modeling.
Change in parental inconsistency, as measured by the Parenting Inconsistency Scale | Baseline, within 1 week post-treatment, 3 months follow-up
  Parenting Inconsistency Scale has 9 items answered on a 5-point Likert scale that ranges from 1 (does not describes me at all) to 5 (describes me completely). The total score can range from 1 to 5, with higher scores indicating a higher level of parental inconsistency.
Change in parental depressive symptoms, as measured by the Patient Health Questionnaire-9 (PHQ-9). | Baseline, within 1 week post-treatment, 3 months follow-up
  The Patient Health Questionnaire-9 is a brief self-report measure used to monitor the severity of depression symptoms. The scale has 9 items answered on a 4-point Likert scale that ranges from 0 (not at all) to 3 (nearly every day). The total score can range from 0 to 27, with higher scores indicating higher levels of depression severity.
Change in parental anxiety symptoms, as measured by the General Anxiety Disorder-7 (GAD-7). | Baseline, within 1 week post-treatment, 3 months follow-up
  The General Anxiety Disorder-7 is a brief self-report measure used to monitor the severity of anxiety symptoms. The scale has 7 items answered on a 4-point Likert scale that ranges from 0 (not at all) to 3 (nearly every day). The total score can range from 0 to 21, with higher scores indicating higher levels of anxiety severity.

OTHER OUTCOMES:
Parents' motivation to participate in the intervention, as measured by the Motivation for Change Rating Scale - Parental Version (MCRS) | Baseline
  The Motivation for Change Rating Scale - Parental Version is a questionnaire developed by the research team for the purpose of assessing parents' motivation for change. The scale has 6 items answered on a 5-point Likert scale that ranges from 0 (nothing) to 4 (very much). The total score can range from 0 to 24, with higher scores indicating higher levels of motivation to change.
Parents' self-efficacy and enjoyment in using the internet and technology | Baseline
  Parents' self-efficacy and enjoyment in using technology will be measured by a questionnaire developed by the research team. The scale has 3 items answered on a 5-point Likert scale that ranges from 0 (nothing) to 4 (very much). The total score can range from 0 to 12, with higher scores indicating higher levels of self-efficacy and enjoyment.
Children's self-efficacy and enjoyment in using the internet and technology | Baseline
  Children's self-efficacy and enjoyment in using technology will be measured by a questionnaire developed by the research team. The scale has 3 items answered on a 5-point Likert scale that ranges from 0 (nothing) to 4 (very much). The total score can range from 0 to 12, with higher scores indicating higher levels of self-efficacy and enjoyment.
Parental beliefs about child anxiety, as measured by the Parental Beliefs About Child Anxiety Questionnaire (PBA-Q) | Baseline
  A brief version of the Parental Beliefs About Child Anxiety Questionnaire will be used to assess parents' anxious reactions to their children's physical symptoms and parents' negative beliefs about their children's experience of anxiety. The brief version has 4 items answered on a 4-point Likert scale that ranges from 0 (completely disagree) to 3 (completely agree). The total score can range from 0 to 12, with higher scores indicating higher levels of parents' negative beliefs about their children's experience of anxiety.
Parents' involvement in therapy, as measured by the Parental Involvement in Therapy Scale (PITS) | within 1 week post-treatment
  The Parental Involvement in Therapy Scale is a four-item scale that asks the clinician to evaluate parents' involvement in the therapy. Items are answered on a 5-point Likert scale that ranges from 0 to 5. The total score can range from 0 to 20, with higher scores indicating higher levels of parents' involvement.
Feasibility of the intervention as measured by adherence | within 1 week post-treatment
  The feasibility of the psychological interventions will be measured through adherence (number of treatment completers).
Feasibility of the intervention as measured by drop-out rates | within 1 week post-treatment
  The feasibility of the psychological interventions will be measured through dropout rates (number of participants that dropped out from the intervention before completing it).
Feasibility of the intervention as measured by the pattern of the online sessions usage | within 1 week post-treatment
  Measured through specific questions (to be developed by the researchers) to assess usability.
Acceptability of the intervention | within 1 week post-treatment
  Measured through specific questions (to be developed by the researchers) to assess acceptability.

CONTACTS AND LOCATIONS:
Overall Officials: Helena Moreira, PhD, Principal Investigator — University of Coimbra
Locations (2):
- Portugal (2):
  - Faculty of Psychology and Educational Sciences, Coimbra
  - Faculty of Psychology, University of Lisbon, Lisbon

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Moreira H, Skvarc D, Gomes-Pereira B, Albuquerque A, Gois AC, Fonseca A, Pereira AM, Caiado B, Paulino B, Santos C, Ehrenreich-May J, Canavarro MC, Saraiva M, Vicente VN, Pereira AI. Study protocol for a randomized controlled trial testing the efficacy of Emotion Detectives In-Out: a blended version of the unified protocol for transdiagnostic treatment of emotional disorders in Portuguese children. BMC Psychol. 2024 Feb 7;12(1):63. doi: 10.1186/s40359-024-01532-z. PMID 38326847